CLINICAL TRIAL: NCT06509867
Title: The Clinical and Patient Morbidity Comparison of De-Epithelialized Gingival Graft With or Without Platelet Rich Fibrin in Multiple Gingival Recessions: A Split-mouth, Randomized Controlled Study
Brief Title: Comparison of De-Epithelialized Gingival Graft With or Without Platelet Rich Fibrin in Multiple Gingival Recessions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Berceste Guler, Assoc Prof, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E.4712136290600/110
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Gingival Recession, Generalized
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: A total of 15 patients were surgically treated with coronally advanced flap (CAF) associated with de-epithelialized gingival graft. Groups were defined as DGG and DGG+PRF:
  DGG Group (n=15): de-epithelialized subepithelial connective tissue grafts + coronally advanced flap DGG+PRF Group (n=15): de-epithelialized subepithelial connective tissue grafts+ L-Platelet Rich Fibrin + Coronally advanced flap
Who Masked: Investigator, Outcomes Assessor
Masking Description: All clinical measurements will be measured and recorded by the blinded researcher. Treatment assignment and surgeries will have been unknown to this examiner. For statistically analysis, groups will be anonymized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Platelet rich fibrin (Experimental): de-epithelialized subepithelial gingival grafts+ L-Platelet Rich Fibrin + Coronally advanced flap
  Interventions: Procedure: DGG+PRF
- de-epithelialized gingival grafts (Active Comparator): de-epithelialized gingival grafts + coronally advanced flap
  Interventions: Procedure: DGG

INTERVENTIONS:
Procedure: DGG+PRF — de-epithelialized subepithelial connective tissue grafts+ L-Platelet Rich Fibrin + Coronally advanced flap
  Other Names: platelet rich fibrin
  Arms: Platelet rich fibrin
Procedure: DGG — de-epithelialized subepithelial connective tissue grafts+ Coronally advanced flap
  Other Names: de-epithelialized gingival graft
  Arms: de-epithelialized gingival grafts

SUMMARY:
The aim of this study is to compare the clinical efficacy and patient reported outcome measures of de-epithelialized gingival graft (DGG) with or without platelet rich fibrin on treatment of multiple adjacent gingival recessions with coronally advanced flap (CAF) technique.

DETAILED DESCRIPTION:
Fifteen patients with split-mouth multiple gingival recessions affecting at least 3 adjacent teeth will be treated with either DGG or DGG+PRF. Recession depth(RD) and width(RW), probing depth(PD), clinical attachment level(CAL), keratinized tissue width (KTW), gingival thickness(GT), and percentage of root coverage (RC%) will be evaluated at 1, 3 and 6 months postoperatively. For patient reported outcome measurements, oral health impact factor-14 (OHIP-14) scores, postoperative pain, bleeding, discomfort and painkiller consumption will be recorded.

A total of 15 patients will surgically treated with coronally advanced flap (CAF) associated with de-epithelialized gingival graft. Groups were defined as DGG and DGG+PRF:

DGG Group (n=15): de-epithelialized subepithelial connective tissue grafts + coronally advanced flap DGG+PRF Group (n=15): de-epithelialized subepithelial connective tissue grafts+ L-Platelet Rich Fibrin + Coronally advanced flap

ELIGIBILITY:
Inclusion criteria of participants were as belows:

Age > 18 years Systemically healthy and non-smoker Full-mouth plaque index and full-mouth gingival index score< 20% No mucogingival surgery experience at operation area No active periodontal disease Patients who have not received orthodontic treatment

Exclusion criteria of participants were as belows:

Pregnancy and lactation Bruxism or occlusal trauma Medical contradictions and for periodontal plastic surgery (i.e. mental disorders) Medication intake

Inclusion criteria of surgical area were as below; Presence of at least three single-rooted teeth (anterior-premolar) with RT1 Class [25] buccal gingival recession defects ≥2 mm in depth Keratinized gingival width<3 mm Sufficient oral hygiene (bleeding on probing <10%, Periodontal Depth<3 mm) Patients without restoration and/or filling in the gingival recession area Absence of non-carious cervical lesions and non-detectable cemento-enamel junction (CEJ) at the defect sites

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
percentage of root coverage | at 6th month
  Percentage of Root Coverage (RC%) were performed with the following formulas. RC%: [(Preoperative RD-Postoperative RD)/ Preoperative RD] x 100.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Faculty of Dentistry, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zucchelli G, Mele M, Stefanini M, Mazzotti C, Marzadori M, Montebugnoli L, de Sanctis M. Patient morbidity and root coverage outcome after subepithelial connective tissue and de-epithelialized grafts: a comparative randomized-controlled clinical trial. J Clin Periodontol. 2010 Aug 1;37(8):728-38. doi: 10.1111/j.1600-051X.2010.01550.x. Epub 2010 Jun 24. PMID 20590963
- [Background] Zucchelli G, Mele M, Mazzotti C, Marzadori M, Montebugnoli L, De Sanctis M. Coronally advanced flap with and without vertical releasing incisions for the treatment of multiple gingival recessions: a comparative controlled randomized clinical trial. J Periodontol. 2009 Jul;80(7):1083-94. doi: 10.1902/jop.2009.090041. PMID 19563288
- [Background] Kuka S, Ipci SD, Cakar G, Yilmaz S. Clinical evaluation of coronally advanced flap with or without platelet-rich fibrin for the treatment of multiple gingival recessions. Clin Oral Investig. 2018 Apr;22(3):1551-1558. doi: 10.1007/s00784-017-2225-9. Epub 2017 Oct 20. PMID 29058084